CLINICAL TRIAL: NCT03592641
Title: A Phase 2 Study of Savolitinib in Subjects With MET Amplified Metastatic Colorectal Cancer
Brief Title: Savolitinib in Treating Patients With MET Amplified Metastatic or Unresectable Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01463; NCI-2018-01463 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-10181; 10181 (Other: Duke University - Duke Cancer Institute LAO); 10181 (Other: CTEP); UM1CA186704 (NIH)
Record Dates: First submitted 2018-07-17; First posted 2018-07-19 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Carcinoma; Metastatic Colon Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Colon Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8; Unresectable Colon Adenocarcinoma; Unresectable Rectal Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (savolitinib) (Experimental): Patients receive savolitinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Savolitinib

INTERVENTIONS:
Drug: Savolitinib — Given PO
  Other Names: AZD 6094; AZD6094; HMPL-504; Volitinib

SUMMARY:
This phase II trial studies how well savolitinib works in treating patients with MET amplified colorectal cancer that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Savolitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the objective response rate (ORR) of savolitinib in patients with MET amplified metastatic colorectal cancer (CRC).

SECONDARY OBJECTIVES:

I. To describe the clinical activity (duration of response, progression free survival [PFS]) of savolitinib in patients with MET amplified metastatic CRC.

II. To describe the toxicities of savolitinib in patients with MET amplified metastatic CRC.

III. To explore the effect of RAS mutation status on response to savolitinib. IV. To explore any correlation between tissue and blood based biomarkers and clinical outcomes.

OUTLINE:

Patients receive savolitinib orally (PO) once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 12 weeks thereafter for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is metastatic and/or unresectable
* Documented wild-type in KRAS and NRAS (codons 12, 13, 59, 61, 117, and 146) and in BRAF codon 600, based on tumor tissue taken from primary or metastatic site prior to anti-EGFR antibody treatment
* At least one site of disease that is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* MET amplification detected by the Guardant360 circulating free deoxyribonucleic acid (cfDNA) screening assay (MET copy number >= 2.2)
* Clinical or radiographic progression on treatments containing a fluoropyrimidine (e.g., 5- fluorouracil or capecitabine), oxaliplatin, irinotecan, and an anti-VEGF monoclonal antibody (bevacizumab, ziv-aflibercept) or anti-VEGFR monoclonal antibody (ramucirumab), and an anti-PD1 monoclonal antibody (nivolumab or pembrolizumab) for patients with microsatellite instability (MSI)-high/mismatch repair (MMR) deficient tumors, or the treatments were not tolerated or contraindicated
* Clinical or radiographic progression on prior anti-EGFR antibody therapy (either panitumumab or cetuximab)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky >= 80%)
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Hemoglobin (Hgb) >= 9 g/dL (no transfusion in the past 2 weeks)
* Platelets >= 100,000/mcL (no transfusion in the past 10 days)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x the institutional upper limit of normal (ULN) with total bilirubin (TBL) =< 1 x ULN OR
* Total bilirubin (TBL) > ULN =<1.5 × ULN with ALT and AST =< 1x ULN
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* International normalization ratio (INR) < 1.5 x ULN and activated partial thromboplastin time (aPTT) < 1.5 x ULN unless patients are receiving therapeutic anticoagulation which affects these parameters
* Females of childbearing potential should be willing to use adequate contraceptive measures, should not be breast feeding, and must have a negative pregnancy test if of childbearing potential or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal is defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments; women under the age of 50 years would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for the institution; or women with documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Male patients with female partner of childbearing potential should be willing to use barrier contraception during the study and for 6 months following discontinuation of study drug
* Ability to swallow and retain oral medications
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g. cytokines or antibodies) within 3 weeks of first dose of study treatment
* Not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from adverse events due to all prior anti-cancer therapies except alopecia, oxaliplatin-related neuropathy, and other non-clinically significant adverse events
* Any other investigational agents within 21 days before the first dose of study treatment
* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered =< 28 days or limited field radiation for palliation =< 7 days prior to starting study drug or has not recovered from side effects of such therapy
* Known brain metastases. (Radiated or resected lesions are permitted, provided the lesions are fully treated and inactive, patient is asymptomatic, and no steroids have been administered for at least 30 days)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to savolitinib
* Prior treatment with a small molecule inhibitor of c-MET or monoclonal antibody against c-MET or HGF
* Any of the following concurrent medication use:

  * Herbal preparations/medications are not allowed throughout the study. These herbal medications include, but are not limited to: St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (dhea), yohimbe, saw palmetto, and ginseng. Patients should stop using these herbal medications 7 days prior to first dose of study drug (three weeks for St. John's wort)
  * Patients receiving or requiring strong inducers or strong inhibitors of CYP3A4, strong inhibitors of CYP1A2, or CYP3A4 substrates which have a narrow therapeutic range within 2 weeks of the first dose of study treatment (3 weeks for St John's wort) will be excluded
  * Concomitant use of drugs that are known to be strong inhibitors of CYP3A4 or CYP1A2 is not permitted during the trial or must be stopped at least 2 weeks prior to receiving the first dose of savolitinib
* Any of the following cardiac disease currently or within the last 6 months:

  * Unstable angina pectoris
  * Congestive heart failure (New York Heart Association [NYHA]) >= grade II
  * Acute myocardial infarction
  * Stroke or transient ischemic attack
* Known hypersensitivity to the active or inactive excipients of AZD6094
* Uncontrolled hypertension (blood pressure [BP] >= 150/95 mmHg despite medical therapy)
* Active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea grade >= 2, and malabsorption syndrome)
* Mean resting correct QT interval (Fridericia's correction formula [QTcF]) > 470 msec for women and > 450 msec for men on screening obtained from 3 electrocardiograms (ECGs)
* Any factors that may increase the risk of QTc prolongation such as chronic hypokalemia not correctable with supplements, congenital or familial long QT syndrome; or family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medications known to prolong QT interval and cause Torsades de Pointes (TdP)
* Any clinically important abnormalities in rhythm, conduction or morphology of resting electrocardiograms (ECGs), e.g. complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec
* Major surgical procedures =< 28 days of beginning study drug or minor surgical procedures =< 7 days. No waiting is required following port-a-cath placement
* Serious underlying medical condition at the time of treatment that would impair the ability of the patient to receive protocol treatment
* Active hepatitis B (positive hepatitis b virus [HBV] surface antigen [HBsAg] result) or hepatitis C (hepatitis C virus [HCV]) infection. Patients with positive HCV antibody are eligible only if the polymerase chain reaction is negative for HCV ribonucleic acid (RNA). Patients with a past or resolved HBV infection are eligible if:

  * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc] OR
  * Positive for HBsAg, but for > 6 months have had normal transaminases and HBV DNA levels between 0-2000 IU/ml (inactive carrier state) and willing to start and maintain antiviral treatment for at least the duration of the study OR
  * HBV DNA levels > 2000 IU/ml but on prophylactic antiviral treatment for the past 3 months and will maintain the antiviral treatment during the study
* Known serious active infection requiring antibiotic, antiviral or antifungal therapy. Human immunodeficiency virus (HIV)-positive patients are eligible only if meeting ALL criteria below:

  * No history of acquired immunodeficiency syndrome (AIDS)-defining conditions
  * Has been on the current highly active antiretroviral therapy (HAART) regimen for the past 3 months and will remain on the same regimen during the study
  * Current HAART regimen has a low potential for drug-drug interaction with the study drug
  * HIV viral load consistently below detectable limit for the past 3 months
  * CD4 count consistently > 200 cells/mm^3 for the past 3 months
* Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years. Patients with stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely (less than 5% probability) to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer
* Psychiatric illness/social situations that would limit compliance with study requirements. Patients with impaired decision-making capacity who have a close caregiver or legal guardian are also eligible with the consent of the caregiver/guardian
* Judgment by the investigator that the patients should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Strickler, Principal Investigator — Duke University - Duke Cancer Institute LAO
Locations (33):
- United States (33):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYU Winthrop Hospital, Mineola, New York
  - Bellevue Hospital Center, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Jia J, Moyer A, Lowe M, Bolch E, Kortmansky J, Cho M, Lenz HJ, Kalyan A, Niedzwiecki D, Strickler JH. A Phase 2 study of Savolitinib in Patients with MET Amplified Metastatic Colorectal Cancer. J Gastrointest Cancer. 2024 Dec 9;56(1):29. doi: 10.1007/s12029-024-01156-x. PMID 39652198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 12 health system organizations within the NCI network. Enrollment was open from 1/30/2019 to 12/30/2021.
Pre-assignment Details: 70 subjects were pre-screened to test for MET amplification. 9 subjects had MET amplification and signed the main consent form. 4 of these subjects were excluded from the trial because they did not meet all eligibility criteria. 5 subjects were enrolled in the treatment portion of the study.
Groups:
- Treatment (Savolitinib): savolitinib 600 mg once daily for weight ≥ 50 kg and 400 mg once daily for weight < 50 kg
Period: Overall Study
Arm/Group | Treatment (Savolitinib)
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Savolitinib)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Objective response rate is calculated as the number of people with a complete or partial response divided by the total number of people treated. Complete response is defined as disappearance of all target lesions. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of treatment until documented progression of disease (up to 4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Savolitinib)
Number analyzed (Participants) | 4
Participants | 0

2. Secondary Outcome: Months of Progression-Free Survival (PFS)
Description: Progression-free survival is defined as the duration of time from start of treatment until clinical or radiographic progression or death, whichever occurs first. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From start of treatment until documented progression of disease (up to 4 months)
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Savolitinib)
Number analyzed (Participants) | 4
months | 2.29 [1.41 to 3.55]

ADVERSE EVENTS:
Time Frame: From start of treatment until 1 month after end of treatment (up to 5 months)
Description: Adverse events were described by grade, frequency, and attribution according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 5.0).
Arm/Group | Treatment (Savolitinib)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Savolitinib) (N=5)
anorexia (Metabolism and nutrition disorders) | 1
dizziness (Nervous system disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
sinus tachycardia (Cardiac disorders) | 1
thromboembolic event (Vascular disorders) | 1
edema limbs (General disorders) | 1
vascular access complication (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Savolitinib) (N=5)
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Blood bicarbonate decreased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 3
Indigestion (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Biliary Obstructions (Hepatobiliary disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Common Cold Symptoms (Infections and infestations) | 1
Stubbed Toe (Injury, poisoning and procedural complications) | 1
LDH Increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Pain (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Serum amylase increased (Investigations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 2
Edema limbs (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT03592641/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT03592641/ICF_001.pdf